CLINICAL TRIAL: NCT04483830
Title: Sulodexide in the Treatment of Early Stages of COVID-19
Brief Title: Suloexide in the Treatment of Early Stages of COVID-19
Acronym: SulES-COVID
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Clinedem (Other)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Principal Investigator, alejandro jose gonzalez ochoa, Vascular and endovascular surgery, Clinedem
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clidm/Vas/2020-05-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-23 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Intervention Model Description: prospective, single centre, randomized, placebo-control trial
Who Masked: Participant
Masking Description: placebo control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Placebo Comparator): patient with the early stages of COVID-19 to received an oral dose of placebo twice a day for 21 days
  Interventions: Drug: Placebo
- group B (Active Comparator): patient in the early stages of COVID-19 to received an oral dose of 500LRU of sulodexide twice a day for 21 days.
  Interventions: Drug: Sulodexide

INTERVENTIONS:
Drug: Sulodexide — an oral dose of 2 capsules each day for 21 days
  Other Names: vessel due f
  Arms: group B
Drug: Placebo — an oral dose of 2 capsules each day for 21 days
  Other Names: vessel due f -placebo
  Arms: group A

SUMMARY:
Problem:

The COVID- 19 pandemic has not only affected our healthcare system, but the impact on the worldwide financial systems and our "normal" way of life is still to be determined.

Although the percentage of patients infected with COVID-19 that need hospital care is low, Its high rate of contagiousness makes the total number of patients in need of hospital care cripple any healthcare system, limiting the space available for other patients in need of critical care, who cannot be admitted or even prefer not to attend the hospital in fear of infection.

Early investigations report an Increase risk of thromboembolic complications, and a systemic inflammatory response not clearly understood. There is a possible vascular endothelial dysfunction due to chronic comorbidities (Hypertension, diabetes, obesity, chronic kidney disease, lung disease) as a risk factor for a more severe presentation.

Justification:

Sulodexide is a two-compound drug, each of them with different endothelial action that can be beneficial in COVID-19 patients.

Glycosaminoglycans: Can help restore venous and arterial endothelial glycocalyx which can downregulate or limit the response to inflammatory molecules, by maintaining the integrity lost in certain chronic diseases (high blood pressure, diabetes).

Heparin compound: It has an antithrombotic effect that could help reduce the incidence of thromboembolic complications, and also add to the anti-inflammatory response due to it anti-thrombin action (similar or a bit less to that of low molecular weight heparin) with less risk of major bleeding.

It's a medication that can be used orally with minimal adverse effects and is less expensive than low molecular weight heparin.

Hypothesis:

We hypothesize that sulodexide instituted early in populations at significant risk and symptomatic patients affected with COVID-19 (shortness of breath, fever, weakness, diarrhoea) and risk factors of diabetes, hypertension, COPD, atherosclerosis, chronic kidney disease, will provide improvement in endothelial integrity, decrease inflammatory responses, and improved clinical outcomes with decreased hospital admission, decrease VTE and arterial complications, morbidity, and mortality.

Objective:

To use sulodexide in patients that have early onset of COVID-19 symptoms to mitigate the progression of the disease process that can allow them to recover at home, and limit the need of hospital care and a more severe clinical manifestation

DETAILED DESCRIPTION:
Objective:

To use sulodexide in patients that have early onset of COVID-19 symptoms to mitigate the progression of the disease process that can allow them to recover at home, and limit the need for hospital care and the more severe manifestation which includes fulminant respiratory failure, acute kidney injury, cardiomyopathy, and thrombosis.

Target study population:

COVID-19 positives in the early but symptomatic stages of the disease (fever, cough, shortness of breath, malaise, diarrhoea, nausea, vomiting, anosmia). High risk of developing a severe presentation of the disease (due to chronic comorbidities).

Research methodology Prospectively, information collection will be carried out in COVID-19 patients, who are in early stages of the disease, defined as a beginning of symptoms of 3 days or less, who attend the CLINEDEM medical unit, located in San Luis Rio Colorado, Sonora, Mexico, in the period from June 15, 2020, to 30 August 2020. Demographic and clinical data will be collected digitally and physically and kept in the clinical record individually the researcher.

This is a clinical, prospective, one-centre, randomized, controlled study. The collaboration of the participants in the protocol will be a minimum of 3 weeks. Selection Period: the time during which candidates will be reviewed, selected, and randomized. Contact will be made with primary health services, both government and private, for a prompt reference of suspected cases, contact with family members of known COVID-19 patients to seek evaluation if developing symptoms, and social media recruitment. Candidates will be evaluated for inclusion criteria by the researcher (or the assigned person), explain the protocol, confirm the availability and/or willingness to participate, the signature of informed consent will be obtained for follow-up and laboratory sampling, from then on patients will be considered inscribed in the clinical trial. The physician (or assigned person) will collect general demographic information, relevant medical history, measurement of patient weight and height for body mass index (BMI) calculation, send to a clinical laboratory that will perform baseline examination blood samples, and COVID-19 testing.

2 groups will be formed: Group A: COVID-19 positive patients with early-stage symptoms who will receive placebo doses of sulodexide. Group B: COVID-19 positive patients with early-stage symptoms receiving doses of sulodexide.

Treatment period: time from when patients initiate the oral dose of sulodexide. Patients in groups A and B will receive the recommended initial stage treatment protocol which consists of rest, measures of home isolation, and use of acetaminophen in case of pain or fever. if the participant is indicated another medicine by their treating physician, it will be recorded in their file, but will not be an elimination criterion.

Group A: will be granted supply for 7 days of placebo medicine in the same packaging and appearance as the original sulodexide. A first follow-up appointment will be scheduled, which will be made according to the participant's preference, either virtually (phone, cell phone, videoconference) or physically with a visit to the patient's home by the researcher or a study collaborator, which will be repeated every 7 days for 21 days, questions will be asked about the general health condition and will report adverse symptoms related to drug intake. During this period, extra visits will be made at the request of the patient or consideration of the investigator. At each visit, symptomatic progression will be asses. At the end of the 21 days, a control blood sample will be carried out including dimer-D and C-reactive protein and the study variables will be analyzed.

In case of need for hospital care, the authorization will be requested from the physician is charged to obtain daily information about the general evolution during the stay, without interfering with the specific treatment protocol. This information will be collected and emptied into a database electronically and physically. Despite being part of the initial informed consent, follow-up authorization will be confirmed during a hospital stay, which can be denied at any time by the patient or family member, in case the participant is not in a position to make decisions. The use of a placebo will be ruled out at that time. Group B: the same protocol as group A + Sulodexide dose of 500 LRU will be added every 12hrs (two capsules).

Measures to prevent or minimize bias: Control group will be receiving a placebo. Randomization will be performed according to the Castor EDU computing program. Only the research leader will be known as randomization allocation.

Premature interruption of the study: The study may be suspended prematurely if significant safety problems are detected, if new scientific knowledge arises, or if other conditions arise that place subjects at undue risk if they continue in the study. The sponsor or the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) or the competent authorities may terminate the study before its scheduled time.

Drug compliance The dates of the first and last intake, as well as any interruption of treatment, if any, will be recorded in the participant's file. The number of tablets dispensed and the number of tablets returned by the participant must be counted by the researcher or a designated person on his/her team and registered. If the participant does not bring back their medication box, the number of tablets taken and the number of days in which the means have been applied will be estimated by the investigator interrogating the participant. If the information is available on an upcoming visit, the data should be corrected. Compliance will be evaluated weekly for the duration of your participation. Compliance shall be calculated based on the relationship between the number of tablets taken and the theoretical number of tablets required by the number of treatment days. If compliance is not satisfactory during the study (e.g. less than 80% or more than 120%), the participant should be questioned to identify the reason for the study.

Universe With a population in the area of San Luis Rio Colorado and its surroundings approximately 1,000,000. 60% in the age range between 20 and 70 years and 55% female sex.

There is difficulty in defining the current number of positive cases given the presence of asymptomatic carriers of the disease, as well as a lack of openness for diagnostic tests in the health sector, limiting an adequate sample calculation required for the study.

A COVID-19 patient has an 80% probability of developing a self-limited presentation that will not warrant hospital care, but in the presence of comorbidities, the risk can increase. This trial is focused on high-risk patients that can develop the need for hospital care given by the calculator risk assessment software, increasing the risk of hospital care in our population to 30-50%. In the severe presentation, the risk of mechanical ventilation can be 20% and a 6.7% mortality rate, however, these data can be modified according to different countries and by the presence of risk factors given by chronic commodities.

In Mexico, as of June 07, 2020, the national mortality rate is reported at 11.8% and in the state of Sonora of 9.7%. In the town of San Luis Rio Colorado, Sonora, of the cases confirmed 37.7% has required hospital management.

Sample size:

The sample size was determined using G*Power 3.1.9.2 program by taking an error type I with a value of 5% (alpha-0.05), a type II error of 20% (beta-0.20) giving a 95% confidence value and a statistical power of 80%. Obtaining a No. 102 participants per group to which 10% was added for possible patient loss/abandonment by defining a total sample of 112 patients per study group.

Statistical analysis The data will be emptied into Excel sheets (Office 360, Microsoft) and transferred to the Statistical Package for Social Sciences (SPSS) version 25 (IBM) operating program for statistical analysis.

The study looks for a superior effect in group B (sulodexide) compared to group A (control), a significant level will be set to 5% (p < 0.05) with a 95% confidence interval.

Descriptive variables will be presented as mean, standard deviation (SD), minimum, maximum for continuous data, and a number of cases and percentages for categorical data. The student t-test and chi-square will be used to compare the differences between the two groups accordingly.

Variable Classification Dependents: the need for hospital care, days needed supplemental oxygen, need for hemodialysis, need for mechanical ventilation, mortality, presence of major bleeding, presence of thromboembolic complications, Serum levels of D- dimer, serum levels of C-reactive protein, serum levels of creatinine.

Independent: Use of sulodexide General precautions of sulodexide: If anticoagulants are used simultaneously, the doses of the anticoagulants should be readjusted.

Restrictions on use during pregnancy and lactation: Although fetal toxicity studies did not show embryo or fetal-toxic effects, use during pregnancy or lactation is not recommended.

Secondary and adverse reactions: Epigastric pain, nausea, vomiting, and skin rash have rarely been reported. Local manifestations have occasionally been reported at the site of redness injection or small bruising. In control group research, the frequency of side effects is similar to placebo.

Adverse Events:

All adverse events and other situations relevant to the safety of participants should be followed and documented completely and accurately to ensure that the sponsor has the information necessary to continuously assess the benefit-risk balance of the Clinical Trial. An adverse event is defined as any unfavourable medical occurrence in a subject participating in a clinical study, whether or not there is a causal relationship with the medicinal product understudy, and/or experimental procedures, which occur or are detected from the date on which the participant signs the consent form, regardless of the study period (e.g. the selection period, they also refer).

Therefore, an adverse event may be:

* Any unwanted signs, including an abnormal finding of an additional examination (laboratory tests, x-rays, ECG, etc.) that is considered clinically relevant by the researcher
* Any symptoms or illnesses not related to the underlying disease.

Ethical and Regulatory Aspects

Helsinki Declaration from the World Medical Association: The Global Medical Association has promulgated the Helsinki Declaration as a proposal for ethical principles for medical research in humans, including research of identifiable human material and information.

According to ethical principles for medical research in human beings, the physician has to protect life, health, dignity, integrity, the right to self-determination, privacy and confidentiality of information; Following this principle, the confidentiality of the information will be maintained the participating patients, only medical and administrative personnel related to the protocol will have access to the clinical record where the patient's name and information are located. For third parties who require access to the data, mainly for the final statistical analysis or collaboration of some information regarding the study, this will be sent, subject to authorization by the principal investigator, but under special coding that replaces the name of the participant and not including personal-work information not related to the study.

ELIGIBILITY:
Inclusion Criteria:

* 3 days or less with clinical COVID-19 symptoms (fever, cough, sour throat, headache, body ache, anosmia, diarrhoea, vomiting).
* sign inform consent.
* >50% risk developing a severe clinical presentation of COVID-19 according to risk calculator

Exclusion Criteria:

* COVID-19 negative test
* known pregnancy
* chronic use of steroid medication
* deep vein thrombosis in the last 6 months
* extended anticoagulation in the last 3 months.
* known allergy to sulodexide.
* severe symptoms that warrant hospital care at initial screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
hospital care | 21 days since start of trial participation
  need for hospital care admission
days of hospital care | 21 days since start of trial participation
  number of total days in hospital care
days of need suplemental oxigen | 21 days since the start of trial participation
  total days in need of supplemental oxigen via facial mask or nasal
serum level of d-dimmer | change betwen basal level and at 14 day follow-up
  total value in ng/dl of d-dimmer
serum level of creatinine | change between basal level ans at 14 day followup
  total value in mg/dl

SECONDARY OUTCOMES:
thromboembolic event | 21 days from start of trial
  presence of a tromboembolic event
need for mechanical ventilation | 21 days from the start of the trial
  the need for the use of endotraqueal tube mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro j Gonzalez-Ochoa, md, Principal Investigator — Clinedem
Locations (1):
- Clinedem, San Luis Río Colorado, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No
individual participant data will be confidential

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208